CLINICAL TRIAL: NCT05305534
Title: Clinical Performance Evaluation Study of the QIAstat-Dx® BCID GN and GPF Plus AMR Panels on Positive Blood Culture and Pure Colony Isolates From Subjects With Signs and Symptoms of Bloodstream Infection
Brief Title: QIAstat-Dx® BCID Plus AMR Panels Clinical Performance Study
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SMF-18-0136-1-001
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Blood Disease
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — positive blood culture clinical samples and pure colony samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: QIAstat-Dx® BCID GN and GPF Plus AMR Panels — The performance of QIAstat-Dx® BCID GN and GPF Plus AMR Panels will be evaluated in comparison with another validated comparator method, using residual specimens of positive blood culture. Pure colonies derived from the residual positive blood culture specimens will also be tested

SUMMARY:
Study for performance evaluation of the QIAstat-Dx® BCID Plus AMR GPF-Panel and the QIAstat Dx® BCID Plus AMR GN-Panel in comparison with other chosen comparator methods

DETAILED DESCRIPTION:
This multicenter study aims to evaluate the performance of QIAstat-Dx® BCID Plus AMR GPF-Panel and the QIAstat Dx® BCID Plus AMR GN-Panel with another validated comparator method.

ELIGIBILITY:
Inclusion Criteria:

* Positive (as identified through Gram stain) blood culture media specimens cultured within bottle types listed in IFU.
* Residual and de-identified specimens.
* Specimen from subject who has not previously been enrolled.
* Fresh prospectively collected specimens tested within 24 hours of initial blood culture bottle positivity.
* Frozen prospectively collected specimens frozen within 24 hours of initial blood culture bottle positivity.
* Minimum 1.5 mL volume available
* In stage 2 - Pure colony isolates of Bacilli, Actinobacteria, fungi (except Fusarium), Enterobacterales, Pseudomondales, Nesseriales, Pasteurellales, Bacterioidales, or Xanthomonadales.

Exclusion Criteria:

* Positive Blood Culture specimens inoculated with a sample type other than Blood (i.e. Paracentesis, or other body fluids)
* Specimens collected off-label from the manufacturer's package insert (e.g., less than the minimum required blood volume was collected).
* Frozen specimens which are unable to be cultured after thawing.
* Specimen from subject previously enrolled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of bloodstream infection
Sampling Method: Probability Sample
Enrollment: 2142 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
PPA | 6 moths
  positive percentage agreement
NPA | 6 moths
  negative percentage agreement

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Principal Investigator — QIAGEN Gaithersburg, Inc
Locations (1):
- QIAGEN, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
all samples are residual and anonymized